CLINICAL TRIAL: NCT03528421
Title: Clinical Study to Evaluate the Safety and Efficacy of IM19 CAR-T Cell Therapy in Patients With Relapsed or Refractory CD19-positive Non-Hodgkin's Lymphoma
Brief Title: Assessment of Safety and Efficacy of IM19 for Relapsed or Refractory NHL Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YMCART201705
Record Dates: First submitted 2018-05-07; First posted 2018-05-17 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-05

CONDITIONS: Non Hodgkin Lymphoma
Keywords: CAR-T
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IM19 CAR-T cells (Experimental): 3*10^5/kg，1*10^6/kg，3*10^6/kg IM19 CAR-T cell.Two days before cell infusion, all patients will be treated with fludarabine and Cyclophosphamide for 3 days
  Interventions: Biological: IM19; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: IM19 — CAR-T cells
Drug: Fludarabine — Two days before cell infusion, all patients will be treated with fludarabine for 3 days
Drug: Cyclophosphamide — Two days before cell infusion, all patients will be treated with Cyclophosphamide for 3 days

SUMMARY:
n this study, approximately 30 patients with relapsed or refractory non-Hodgkin's lymphoma (NHL) were recruited for a single reinfusion of IM19-CD28 and IM19-41BB CAR-T cells. Assess the safety, tolerability of treatment, and initially observe the efficacy.

DETAILED DESCRIPTION:
1. Dose-escalation:Patients entered the IM19-41BB or IM19-CD28 group and performed dose escalation studies in three dose groups.
2. According to the results of the previous dose escalation study, select one dose to continue the enrollment of 6 patients for extended studies.

ELIGIBILITY:
Inclusion criteria:

1. Relapsed or refractory CD19-positive non-Hodgkin lymphoma (NHL) patients. 1 Diffuse large B lymphoma (DLBCL), follicular lymphoma (FL), primary mediastinal B-cell lymphoma (PMBCL) patients meet one of the following conditions: I Patients who have relapsed or are refractory after at least 2 previous treatments; II Patients who have relapsed after transplantation. 2 Patients with relapsed or refractory mantle cell lymphoma after at least one treatment.
2. Patients must have evaluable disease evidence;
3. Age ≥ 18 years old;
4. The expected life span is more than 3 months;
5. ECOG score 0-2 points (see Attachment 2);
6. Women of childbearing age have a negative blood pregnancy test before the start of the trial and agree to have effective contraceptive measures during the trial until the last follow-up;
7. Those who voluntarily participate in the trial and sign the informed consent.

Exclusion criteria:

1. Patients with high-risk organ involvement: tumors invade one of the central nervous system, gastrointestinal tract, lungs, pericardium, and large vessels;
2. Those who have a graft-versus-host response and need to use immunosuppressive drugs; or who have a disease of the autoimmune system;
3. Use chemotherapy or radiotherapy within 3 days before the blood collection period;
4. Those who have used systemic steroids within the 5 days prior to the blood sampling period (except recently or currently using inhaled steroids);
5. Use stimulating bone marrow hematopoietic cells to produce drugs (whitening needles, etc.) within 5 days before the blood collection period;
6. Those who have previously used any gene therapy products;
7. History of epilepsy or other diseases of the central nervous system;
8. New York Heart Association (NYHA) class III or above (see Annex 3);
9. creatinine> 1.5 times the upper limit of normal or ALT / AST> 3 times the upper limit of normal or bilirubin> 2 times the normal upper limit;
10. active Hepatitis B or Hepatitis C virus, HIV or other untreated active infections;
11. pregnant or lactating women;
12. suffer from other uncontrolled diseases that the researcher considers inappropriate;
13. Any condition that the investigator believes may increase the subject's risk or interfere with the test results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-05-22 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | 2 years
  >= Grade 3 signs/symptoms,laboratory toxicities,and clinical events that are possibly,likely,or definitely related to study treatment Adverse events assessed according to NCI-CTCAE v4.0 criteria 2.

SECONDARY OUTCOMES:
Overall response rate | 2 years
  (1) a morphologic complete response (CR) or (2) a complete response with incomplete recovery of counts (CRi) (based on NCCN guidelines (National Comprehensive Cancer Network (NCCN), 2014)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Ying Z, He T, Wang X, Zheng W, Lin N, Tu M, Xie Y, Ping L, Zhang C, Liu W, Deng L, Wu M, Feng F, Leng X, Du T, Qi F, Hu X, Ding Y, Lu XA, Song Y, Zhu J. Distribution of chimeric antigen receptor-modified T cells against CD19 in B-cell malignancies. BMC Cancer. 2021 Feb 25;21(1):198. doi: 10.1186/s12885-021-07934-1. PMID 33632155